CLINICAL TRIAL: NCT02460419
Title: Maintenance Capecitabine Plus Best Supportive Care Versus Best Supportive Care for Metastatic Nasopharyngeal Carcinoma: a Multicenter, Randomised, Phase 3 Study.
Brief Title: Maintenance Capecitabine Plus Best Supportive Care Versus Best Supportive Care for Metastatic Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other)
Responsible Party: Principal Investigator, XIANG YANQUN, MD,PhD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015029
Record Dates: First submitted 2015-05-23; First posted 2015-06-02 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; metastasis; capecitabine
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Neoplasm Metastasis | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- maintenance capecitabine (Experimental): maintenance capecitabine plus best supportive care(BSC)
  Interventions: Drug: capecitabine; Other: Best supportive care (BSC)
- best supportive care (Other): Best supportive care and following-up every 6-8 weeks
  Interventions: Other: Best supportive care (BSC)

INTERVENTIONS:
Drug: capecitabine — capecitabine 1250mg/m2 bid, oral, for 14 days, every 3 weeks. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Xeloda
  Arms: maintenance capecitabine
Other: Best supportive care (BSC) — Best supportive care and following-up every 6-8 weeks

SUMMARY:
This multicenter, randomised, phase 3 study is to evaluate the survival benefit of maintenance capecitabine plus best supportive care versus best supportive care for metastatic nasopharyngeal carcinoma patients after disease controlled with TPC palliative chemotherapy.

DETAILED DESCRIPTION:
Firstly diagnosed metastatic nasopharyngeal carcinoma patients will receive 4-6 cycles of palliative chemotherapy with taxol,cisplatin and capecitabine. After disease controlled, they will be randomly assigned to maintenance capecitabine plus best supportive care(BSC) or BSC alone. The primary end point is progression-free survival, the secondary end points are overall survival, duration of response, objective response rate, adverse effects and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Firstly diagnosed metastatic nasopharyngeal carcinoma patients
* Disease controlled after 4-6 cycles of palliative chemotherapy with taxol,cisplatin and capecitabine
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Life expectation at least 12 weeks
* No systemic chemotherapy within 6 months, except for induction chemotherapy or concurrent chemotherapy
* With at least one measurable lesion
* Enough blood test
* Signed informed consent

Exclusion Criteria:

* Sever heart disease
* HIV infection
* Sever infection
* Brain metastasis, except received radical therapy 6 months ago and stable in 4 weeks
* Allogeneic organ transplantation
* Malignancy other than nasopharyngeal carcinoma, except:cervical carcinoma in situ, cured basal cell carcinoma,bladder cancer of Ta,Tis or T1, or any cured cancer for at least 3 years
* Pregnancy or breast feeding
* Difficulty in swallowing
* Received other test drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-04; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
progression-free survival | up to 6 years
  the time from randomization to the progression of disease

SECONDARY OUTCOMES:
overall survival | up to 6 years
  the time from randomization to death
duration of response | up to 6 years
  the time from the date of the first cycle of chemotherapy to the progression of disease
objective response rate | up to 6 years
  CR, PR and SD rate
adverse effects | up to 6 years
  chemotherapy side effects
quality of life of the patients during the Maintenance Capecitabine and/or Best Supportive Care | up to 6 years
  evaluate with FACT-H&N every 3 months after randomiztion

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Guo, MD, Study Chair — Sun Yat-sen University
Locations (1):
- SunYat-senU, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Jin Y, Shi YX, Cai XY, Xia XY, Cai YC, Cao Y, Zhang WD, Hu WH, Jiang WQ. Comparison of five cisplatin-based regimens frequently used as the first-line protocols in metastatic nasopharyngeal carcinoma. J Cancer Res Clin Oncol. 2012 Oct;138(10):1717-25. doi: 10.1007/s00432-012-1219-x. Epub 2012 Jun 10. PMID 22684794
- [Background] Chua DT, Yiu HH, Seetalarom K, Ng AW, Kurnianda J, Shotelersuk K, Krishnan G, Hong RL, Yang MH, Wang CH, Sze WK, Ng WT. Phase II trial of capecitabine plus cisplatin as first-line therapy in patients with metastatic nasopharyngeal cancer. Head Neck. 2012 Sep;34(9):1225-30. doi: 10.1002/hed.21884. Epub 2011 Nov 11. PMID 22076785
- [Background] Leong SS, Wee J, Rajan S, Toh CK, Lim WT, Hee SW, Tay MH, Poon D, Tan EH. Triplet combination of gemcitabine, paclitaxel, and carboplatin followed by maintenance 5-fluorouracil and folinic acid in patients with metastatic nasopharyngeal carcinoma. Cancer. 2008 Sep 15;113(6):1332-7. doi: 10.1002/cncr.23687. PMID 18615622
- [Derived] Han J, Lan X, Tian K, Shen X, He J, Chen N. Cost-effectiveness analysis of capecitabine maintenance therapy plus best supportive care vs. best supportive care alone as first-line treatment of newly diagnosed metastatic nasopharyngeal carcinoma. Front Public Health. 2023 Jan 26;10:1086393. doi: 10.3389/fpubh.2022.1086393. eCollection 2022. PMID 36777769
- [Derived] Liu GY, Li WZ, Wang DS, Liang H, Lv X, Ye YF, Zhao C, Ke LR, Lv SH, Lu N, Bei WX, Cai ZC, Chen X, Liang CX, Guo X, Xia WX, Xiang YQ. Effect of Capecitabine Maintenance Therapy Plus Best Supportive Care vs Best Supportive Care Alone on Progression-Free Survival Among Patients With Newly Diagnosed Metastatic Nasopharyngeal Carcinoma Who Had Received Induction Chemotherapy: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2022 Apr 1;8(4):553-561. doi: 10.1001/jamaoncol.2021.7366. PMID 35175316